CLINICAL TRIAL: NCT02607930
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of GS-9883/Emtricitabine/Tenofovir Alafenamide Versus Abacavir/Dolutegravir/Lamivudine in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Study to Evaluate the Safety and Efficacy of Bictegravir/Emtricitabine/Tenofovir Alafenamide Versus Abacavir/Dolutegravir/Lamivudine in Human Immunodeficiency Virus-1 (HIV-1) Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-380-1489; 2015-004024-54 (EudraCT Number)
Record Dates: First submitted 2015-11-10; First posted 2015-11-18 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: HIV-1 Infection
Keywords: HIV
MeSH Terms: interventions — abacavir, dolutegravir, and lamivudine drug combination; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- B/F/TAF (Experimental): B/F/TAF + ABC/DTG/3TC placebo administered without regard to food for at least 144 weeks.
  Interventions: Drug: B/F/TAF; Drug: ABC/DTG/3TC Placebo
- ABC/DTG/3TC (Active Comparator): ABC/DTG/3TC + B/F/TAF placebo administered without regard to food for at least 144 weeks.
  Interventions: Drug: ABC/DTG/3TC; Drug: B/F/TAF Placebo
- Open-label Phase B/F/TAF to B/F/TAF (Experimental): After Week 144, participants will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants will be given the option to receive open-label (OL) B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF is not commercially available will be given the option to continue OL B/F/TAF until the product becomes accessible through an access program or until Gilead elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: B/F/TAF
- Open-label Phase ABC/DTG/3TC to B/F/TAF (Experimental): After Week 144, participants will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants will be given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF is not commercially available will be given the option to continue OL B/F/TAF until the product becomes accessible through an access program or until Gilead elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: ABC/DTG/3TC — 600/50/300 milligrams (mg) tablets administered orally, once daily
  Other Names: Triumeq®
  Arms: ABC/DTG/3TC
Drug: B/F/TAF — 50/200/25 mg tablets administered orally, once daily, without regard to food
  Other Names: GS-9883/F/TAF; Biktarvy®
  Arms: B/F/TAF; Open-label Phase ABC/DTG/3TC to B/F/TAF; Open-label Phase B/F/TAF to B/F/TAF
Drug: ABC/DTG/3TC Placebo — Tablets administered orally, once daily
  Arms: B/F/TAF
Drug: B/F/TAF Placebo — Tablets administered orally, once daily
  Arms: ABC/DTG/3TC

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a fixed dose combination (FDC) containing bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) versus a FDC containing abacavir/dolutegravir/lamivudine (ABC/DTG/3TC) in HIV-1 infected, antiretroviral treatment naive-adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Antiretroviral treatment naive (≤ 10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection) except the use for pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP), up to one month prior to screening
* Plasma HIV-1 ribonucleic acid (RNA) levels ≥ 500 copies per milliliter (mL) at screening
* Adequate renal function: Estimated glomerular filtration rate ≥ 50 milliliter per minute (mL/min) (≥ 0.83 milliliter per second [mL/sec]) according to the Cockcroft-Gault formula
* Negative screening test for human leukocyte antigen (HLA) -B x 5701 allele provided by Gilead Sciences

Key Exclusion Criteria:

* An opportunistic illness indicative of stage 3 HIV diagnosed within the 30 days prior to screening (refer to study protocol)
* Decompensated cirrhosis (e.g, ascites, encephalopathy, or variceal bleeding)
* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
* Females who are pregnant (as confirmed by positive serum pregnancy test)
* Females who are breastfeeding
* Chronic Hepatitis B Virus (HBV) infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (121):
- United States (78):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - Pueblo Family Physicians, Phoenix, Arizona
  - Kaiser Permanente Medical Center, Los Angeles, California
  - Ruane Clinical Research Group, Inc., Los Angeles, California
  - Anthony Martin Mills MD A Medical Corporation, DBA Mills Clinical Research, Los Angeles, California
  - Alameda Health System- Highland Hospital, Oakland, California
  - University of California Davis, Sacramento, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - Kaiser Permanente, San Leandro, California
  - The Lundquist Institute for BioMedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Apex Research, Denver, Colorado
  - Whitman-Walker Institute, Washington D.C., District of Columbia
  - Providence Hospital - DC, Washington D.C., District of Columbia
  - Capital Medical Associates, Washington D.C., District of Columbia
  - Medical Faculty Associates, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Gary J. Richmond, M.D., P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - AHF Kinder Medical Group, Miami, Florida
  - Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - AIDS Healthcare Foundation-Miami Beach, Pensacola, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - AIDS Research and Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Infectious Disease Group PC, Atlanta, Georgia
  - Aids Research Consortium of Atlanta Inc, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Baystate Medical Center, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Kansas City CARE Clinic, Kansas City, Missouri
  - Southampton Clinical Research Group, Inc., St Louis, Missouri
  - Southampton Healthcare Inc, St Louis, Missouri
  - Prime healthcare services - St Michael's LLC d/b/a Saint Michael's medical center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Santa Fe, New Mexico
  - Upstate Infectious Disease Associates, Albany, New York
  - Evergreen Health, Buffalo, New York
  - North Shore University Hospital-(Manhasset), Manhasset, New York
  - Bronx Care, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Aids Research Consortium of Atlanta Inc, Chapel Hill, North Carolina
  - ID Consultants PA, Charlotte, North Carolina
  - Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest Baptist Medical Center - PPDS, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Research Institute, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Medical University of South Carolina PPDS, Columbia, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - Saint Hope Foundation Inc, Bellaire, Texas
  - AIDS Arms Inc, Dallas, Texas
  - UT Southwestern Clinical Trials Office, Dallas, Texas
  - North Texas Infectious Diseases Consultants PA, Dallas, Texas
  - Fort Worth, Texas
  - Therapeutic Concepts, Houston, Texas
  - Gordon E Crofoot MD PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - Diagnostic Clinic of Longview Center For Clinical Research (DCOL), Longview, Texas
  - Peter Shalit MD, Seattle, Washington
  - Multicare Rockwood HIV Critical Care Clinic, Spokane, Washington
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
- Canada (8):
  - Clinique Medicale L'actuel, Montreal
  - McGill University Health Center, Montreal
  - Clinique OPUS Inc, Montreal
  - Ottawa Hospital, Ottawa
  - Sunnybrook Health Sciences Centre, Toronto
  - Maple Leaf Research, Toronto
  - Spectrum Health Care, Vancouver
  - Winnipeg Regional Health Authority, Winnipeg
- Instituto Dominicano de Estudios Virologicos IDEV, Santo Domingo, Dominican Republic
- France (6):
  - Hôpital de La Croix Rousse, Lyon
  - CHU de Nice Archet I, Nice
  - Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Groupe Hospitalier Bichat Claude Bernard, Tourcoing
- Germany (3):
  - zibp Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH, Berlin
  - Universitätsklinikum Bonn, Bonn
  - ICH Study Center, Hamburg
- Italy (3):
  - ASST Papa Giovanni XXIII - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
  - Istituto Nazionale Malattie Infettive Lazzaro Spallanzani IRCCS, Roma
- Puerto Rico (2):
  - Hope Clinical Research, San Juan
  - University of Puerto Rico, San Juan
- Spain (10):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Bellvitge, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo
- United Kingdom (8):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Barts Health NHS Trust, Royal London Hospital, Ambrose King Centre, London
  - Royal Free London NHS Foundation Trust, London
  - Kings College Hospital, London
  - Chelsea and Westminster NHS Trust, London
  - Mortimer Market Centre, London
  - North Manchester General Hospital - PPDS, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Result] Wohl D, Clarke A, Maggiolo F, Garner W, Laouri M, Martin H, Quirk E. Patient-Reported Symptoms Over 48 Weeks Among Participants in Randomized, Double-Blind, Phase III Non-inferiority Trials of Adults with HIV on Co-formulated Bictegravir, Emtricitabine, and Tenofovir Alafenamide versus Co-formulated Abacavir, Dolutegravir, and Lamivudine. Patient. 2018 Oct;11(5):561-573. doi: 10.1007/s40271-018-0322-8. PMID 29956087
- [Result] Wohl DA, Yazdanpanah Y, Baumgarten A, Clarke A, Thompson MA, Brinson C, Hagins D, Ramgopal MN, Antinori A, Wei X, Acosta R, Collins SE, Brainard D, Martin H. Bictegravir combined with emtricitabine and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection: week 96 results from a randomised, double-blind, multicentre, phase 3, non-inferiority trial. Lancet HIV. 2019 Jun;6(6):e355-e363. doi: 10.1016/S2352-3018(19)30077-3. Epub 2019 May 5. PMID 31068270
- [Result] Acosta RK, Willkom M, Martin R, Chang S, Wei X, Garner W, Lutz J, Majeed S, SenGupta D, Martin H, Quirk E, White KL. Resistance Analysis of Bictegravir-Emtricitabine-Tenofovir Alafenamide in HIV-1 Treatment-Naive Patients through 48 Weeks. Antimicrob Agents Chemother. 2019 Apr 25;63(5):e02533-18. doi: 10.1128/AAC.02533-18. Print 2019 May. PMID 30803969
- [Result] Acosta R, Willkom M, Martin R, Chang S, Liu X, Hedskog C, et al. Low-frequency resistance variants in art-naïve participants do not affect bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) triple therapy outcome. [Poster MOPEB242]. 10th IAS Conference on HIV Science (IAS 2019); 2019 July 21-24; Mexico City, Mexico.
- [Result] Acosta R, White K, Garner W, Wei X, Andreatta K, Willkom M, et al. HIV-1 subtype (B or non-B) had no impact on the efficacy of B/F/TAF or resistance development in five phase 3 treatment-naïve or switch studies. [Poster THPEB077]. 22nd International AIDS Conference; 2018 July 23-27; Amsterdam, Netherlands.
- [Result] White K, Kulkarni R, Willkom M, Martin R, Chang S, Wei X, et al. Pooled week 48 efficacy and baseline resistance: B/F/TAF in treatment-naive patients. [Poster 532]. Conference on Retroviruses and Opportunistic Infections; 2018 March 4-7; Boston, USA.
- [Result] Gallant J, Lazzarin A, Mills A, Orkin C, Podzamczer D, Tebas P, Girard PM, Brar I, Daar ES, Wohl D, Rockstroh J, Wei X, Custodio J, White K, Martin H, Cheng A, Quirk E. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection (GS-US-380-1489): a double-blind, multicentre, phase 3, randomised controlled non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2063-2072. doi: 10.1016/S0140-6736(17)32299-7. Epub 2017 Aug 31. PMID 28867497
- [Result] Orkin C, DeJesus E, Sax PE, Arribas JR, Gupta SK, Martorell C, Stephens JL, Stellbrink HJ, Wohl D, Maggiolo F, Thompson MA, Podzamczer D, Hagins D, Flamm JA, Brinson C, Clarke A, Huang H, Acosta R, Brainard DM, Collins SE, Martin H; GS-US-380-1489; GS-US-380-1490 study investigators. Fixed-dose combination bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir-containing regimens for initial treatment of HIV-1 infection: week 144 results from two randomised, double-blind, multicentre, phase 3, non-inferiority trials. Lancet HIV. 2020 Jun;7(6):e389-e400. doi: 10.1016/S2352-3018(20)30099-0. PMID 32504574
- [Result] Acosta R, Andreatta K, D'Antoni M, Collins S, Martin H, White K. HIV Viral Blips in Adults Treated with INSTI-Based Regimens Through 144 Weeks. [Poster 540]. Conference on Retroviruses and Opportunistic Infections 2020 (CROI 2020); 2020 March 8-11; Boston, Massachusetts.
- [Result] Mills A, Gupta SK, Brinson C, Workowski K, Clarke A, Antinori A, Stephens JL, et al. 144-Week Efficacy and Safety of B/F/TAF in Treatment-Naive Adults Age ≥50 Years. [Poster 477]. Conference on Retroviruses and Opportunistic Infections 2020 (CROI 2020); 2020 March 8-11; Boston, Massachusetts.
- [Result] Ramgopal M, Maggiolo F, Ward D, Leboucche B, Rizzardini G, Molina JM, et al. Pooled Analysis of 4 International Trials of Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF) in Adults Aged ≥ 65 Years Demonstrating Safety and Efficacy: Week 48 Results. [Oral OAB0403].AIDS 2020; 2020 July 6-10; Virtual.
- [Result] Acosta R, Andreatta K, D'Antoni M, Collins S, Martin H, White K. Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) shows high efficacy in clinical study participants infected with HIV-1 subtype F. [Poster P124]. HIV Drug Therapy 2020 (HIV Glasgow 2020); 2020 October 5-8; Glasgow, United Kingdom.
- [Result] Workowski K, Orkin C, Sax P, Hagins D, Koenig E, Stephens JL, et al. Four-Year Outcomes of B/F/TAF in Treatment-Naïve Adults [Poster 415]. Conference on Retroviruses and Opportunistic Infections 2021 (CROI 2021); 2021 June 3-November 3; Virtual.
- [Result] Acosta RK, Chen GQ, Chang S, Martin R, Wang X, Huang H, Brainard D, Collins SE, Martin H, White KL. Three-year study of pre-existing drug resistance substitutions and efficacy of bictegravir/emtricitabine/tenofovir alafenamide in HIV-1 treatment-naive participants. J Antimicrob Chemother. 2021 Jul 15;76(8):2153-2157. doi: 10.1093/jac/dkab115. PMID 33880558
- [Result] Arribas J, Orkin C, Maggiolo F, Antinori A, Lazzarin A, Yasdanpanah, et al. Long-term Analysis of B/F/TAF in Treatment-Naïve Adults Living With HIV Through Four Years of Follow-up. [PEB151]. 11th IAS Conference on HIV Science (IAS 2021); 2021 July 18-21; Virtual.
- [Result] Acosta R, Chen G, Qin L, Wang X, Huang H, Hindman J, et al. Achievement of Undetectable HIV-1 RNA in the B/F/TAF Treatment-Naïve Clinical Trials. [Poster PEB150]. 11th IAS Conference on HIV Science (IAS 2021); 2021 July 18-21; Virtual.
- [Result] Acosta R, Chen G, Chang S, Martin R, Wang X, Huang H, et al. HIV with Transmitted Drug Resistance Is Durably Suppressed by B/F/TAF at Week 144. [Poster 430]. Conference on Retroviruses and Opportunistic Infections 2021 (CROI 2021); 2021 June 3-November 3; Virtual.
- [Result] Acosta R, Chen G, Huang H, Liu H, White K. Unreturned Pill Bottles in the 1489 and 1490 Clinical Trials: An Important Measure of Poor Adherence That Is Often Ignored in Pill Count Calculations. [Poster 902]. IDWeek 2021; 2021 September 29-October 3; Virtual.
- [Result] Daar E, Orkin C, Sax P, Stephens J, Koenig E, Clarke A, et al. Incidence of Metabolic Complications Among Treatment-naïve Adults Living With HIV-1 Randomized to B/F/TAF, DTG/ABC/3TC or DTG + F/TAF After 3 Years. [Oral 69]. IDWeek 2021; 2021 September 29-October 3; Virtual.
- [Result] Pozniak A, et al. Outcomes 48 Weeks After Switching From DTG/ABC/3TC or DTG + F/TAF to B/F/TAF. [PE2/68]. 18th European AIDS Conference (EAC 2021), 2021 October 27-30; London, United Kingdom.
- [Derived] Sax PE, Hindman JT, Martin H, Wohl D. Two 5-year studies of bictegravir/emtricitabine/tenofovir alafenamide in people with HIV: a plain-language summary. Future Microbiol. 2024;19(14):1185-1193. doi: 10.1080/17460913.2024.2372231. Epub 2024 Sep 4. PMID 39229805
- [Derived] Orkin C, Antinori A, Rockstroh JK, Moreno-Guillen S, Martorell CT, Molina JM, Lazzarin A, Maggiolo F, Yazdanpanah Y, Andreatta K, Huang H, Hindman JT, Martin H, Pozniak A. Switch to bictegravir/emtricitabine/tenofovir alafenamide from dolutegravir-based therapy. AIDS. 2024 Jun 1;38(7):983-991. doi: 10.1097/QAD.0000000000003865. Epub 2024 Feb 21. PMID 38349226
- [Derived] Sax PE, Arribas JR, Orkin C, Lazzarin A, Pozniak A, DeJesus E, Maggiolo F, Stellbrink HJ, Yazdanpanah Y, Acosta R, Huang H, Hindman JT, Martin H, Baeten JM, Wohl D; GS-US-380-1489 and GS-US-380-1490 study investigators. Bictegravir/emtricitabine/tenofovir alafenamide as initial treatment for HIV-1: five-year follow-up from two randomized trials. EClinicalMedicine. 2023 May 11;59:101991. doi: 10.1016/j.eclinm.2023.101991. eCollection 2023 May. PMID 37200995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in Europe, Dominican Republic, and North America. The first participant was screened on 13 November 2015. The last study visit occurred on 02 July 2021.
Pre-assignment Details: 739 participants were screened.
Groups:
- B/F/TAF: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) tablets fixed-dose combination (FDC) + abacavir (ABC)/dolutegravir (DTG)/lamivudine (3TC) (ABC/DTG/3TC) placebo orally once daily for at least 144 weeks, without regard to food.
- ABC/DTG/3TC: Abacavir/dolutegravir/lamivudine (ABC/DTG/3TC) (600/50/300 mg) FDC tablet + B/F/TAF placebo orally once daily for 144 weeks, without regard to food.
- B/F/TAF to B/F/TAF: After Week 144, participants continued to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive open-label (OL) B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
- ABC/DTG/3TC to B/F/TAF: After Week 144, participants continued to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
Period: Double-Blinded Treatment Phase
Arm/Group | B/F/TAF | ABC/DTG/3TC | B/F/TAF to B/F/TAF | ABC/DTG/3TC to B/F/TAF
Started | 316 | 315 | 0 | 0
Completed | 262 | 262 | 0 | 0
Not Completed | 54 | 53 | 0 | 0
Not completed — Lost to Follow-up | 25 | 19 | 0 | 0
Not completed — Withdrew consent | 14 | 18 | 0 | 0
Not completed — Investigator's discretion | 6 | 3 | 0 | 0
Not completed — Non-compliance with study drug | 3 | 5 | 0 | 0
Not completed — Protocol Violation | 2 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0
Not completed — Randomized but never treated | 2 | 0 | 0 | 0
Period: Open-Label B/F/TAF Extension Phase
Arm/Group | B/F/TAF | ABC/DTG/3TC | B/F/TAF to B/F/TAF | ABC/DTG/3TC to B/F/TAF
Started | 0 (At the End of Blinded Treatment Visit, participants were given the option to receive B/F/TAF FDC in an OL extension phase for up to 96 weeks.) | 0 (At the End of Blinded Treatment Visit, participants were given the option to receive B/F/TAF FDC in an OL extension phase for up to 96 weeks.) | 252 (10 participants from B/F/TAF arm did not enter the Open-Label Extension Phase.) | 254 (8 participants from the ABC/DTG/3TC arm did not enter the Open-Label Extension Phase.)
Completed | 0 | 0 | 218 | 221
Not Completed | 0 | 0 | 34 | 33
Not completed — Lost to Follow-up | 0 | 0 | 15 | 10
Not completed — Withdrew consent | 0 | 0 | 10 | 13
Not completed — Investigator's discretion | 0 | 0 | 2 | 5
Not completed — Adverse Event | 0 | 0 | 4 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- B/F/TAF: Blinded Phase: B/F/TAF (50/200/25 mg) FDC tablet + ABC/DTG/3TC placebo orally once daily for at least 144 weeks, without regard to food
  Open-Label Extension Phase: After Week 144, participants will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants will be given the option to receive open-label (OL) B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF is not commercially available will be given the option to continue OL B/F/TAF until the product becomes accessible through an access program or until Gilead elects to discontinue the study in that country, whichever occurs first.
- ABC/DTG/3TC: Blinded Phase: ABC/DTG/3TC (600/50/300 mg) FDC tablet + B/F/TAF placebo orally once daily for at least 144 weeks, without regard to food
  Open-Label Extension Phase: After Week 144, participants will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants will be given the option to receive open-label (OL) B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF is not commercially available will be given the option to continue OL B/F/TAF until the product becomes accessible through an access program or until Gilead elects to discontinue the study in that country, whichever occurs first.
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | ABC/DTG/3TC | Total
Number analyzed (Participants) | 314 | 315 | 629
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.9) | 34 (10.8) | 34 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 285 | 282 | 567
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = Local regulators did not allow collection of race.
  Participants
    Race: American Indian or Alaska Native | 2 | 4 | 6
    Race: Asian | 6 | 10 | 16
    Race: Black | 114 | 112 | 226
    Race: Native Hawaiian or Pacific Islander | 1 | 2 | 3
    Race: White | 180 | 179 | 359
    Race: Other | 9 | 8 | 17
    Race: Not Permitted | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = Local regulators did not allow collection of ethnicity.
  Participants
    Ethnicity: Hispanic or Latino | 72 | 65 | 137
    Ethnicity: Not Hispanic or Latino | 240 | 249 | 489
    Ethnicity: Not Permitted | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 18 | 15 | 33
  Belgium | 4 | 2 | 6
  United States | 228 | 233 | 461
  Dominican Republic | 2 | 1 | 3
  Italy | 7 | 11 | 18
  United Kingdom | 20 | 11 | 31
  France | 11 | 10 | 21
  Germany | 4 | 9 | 13
  Spain | 20 | 23 | 43
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.41 (0.647) | 4.42 (0.685) | 4.42 (0.665)
HIV-1 RNA Categories [Count of Participants; unit: Participants]
  ≤ 100,000 copies/mL | 261 | 265 | 526
  > 100,000 ≤ 400,000 copies/mL | 45 | 38 | 83
  > 400,000 copies/mL | 8 | 12 | 20
CD4 Cell Count [Mean (Standard Deviation); unit: Cells/µL] | 453 (220.8) | 476 (231.4) | 464 (226.3)
CD4 Cell Count Categories [Count of Participants; unit: Participants]
  < 50 Cells/µL | 7 | 10 | 17
  ≥ 50 to < 200 Cells/µL | 29 | 22 | 51
  ≥ 200 to < 350 Cells/µL | 69 | 58 | 127
  ≥ 350 to < 500 Cells/µL | 87 | 91 | 178
  ≥ 500 Cells/µL | 122 | 134 | 256
Hip Bone Mineral Density (BMD) [Mean (Standard Deviation); unit: g/cm^2] — Population: The Hip Dual-energy X-ray Absorptiometry (DXA) Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, and had non-missing values for baseline hip BMD.
  g/cm^2
    number analyzed (Participants) | 300 | 297 | 597
    (all) | 1.048 (0.1572) | 1.057 (0.1520) | 1.052 (0.1546)
Spine BMD [Mean (Standard Deviation); unit: g/cm^2] — Population: The Spine DXA Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, and had nonmissing values for baseline spine BMD.
  g/cm^2
    number analyzed (Participants) | 304 | 299 | 603
    (all) | 1.139 (0.1847) | 1.142 (0.1713) | 1.140 (0.1780)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- B/F/TAF: Blinded Phase: B/F/TAF (50/200/25 mg) FDC tablet + ABC/DTG/3TC placebo orally once daily for at least 144 weeks, without regard to food.
- ABC/DTG/3TC: Blinded Phase: ABC/DTG/3TC (600/50/300 mg) FDC tablet + B/F/TAF placebo orally once daily for at least 144 weeks, without regard to food.
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 314 | 315
percentage of participants | 92.4 | 93.0
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Non-Inferiority — A sample of approximately 600 participants randomized 1:1 achieves at least 95% power using a non-inferiority margin of 12% assuming a response rate in both groups of 91% (Reference Genvoya studies) and a one-sided alpha level of 0.025; Difference in Percentages = -0.6, 95.002% CI 2-sided [-4.8 to 3.6] — Differences in percentages of participants between groups and their 95.002% CIs were calculated based on Mantel-Haenszel (MH) proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)
Statistical Analysis 2: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Superiority; p = 0.78, Cochran-Mantel-Haenszel; p-value was calculated from CMH test stratified by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)

2. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 96 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 314 | 315
percentage of participants | 87.9 | 89.8
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; Difference in Percentages = -1.9, 95% CI 2-sided [-6.9 to 3.1] — Differences in percentages of participants between groups and their 95% CIs were calculated based on Mantel-Haenszel (MH) proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)
Statistical Analysis 2: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.45, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 144 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 144 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 144
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 314 | 315
percentage of participants | 81.5 | 84.1
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; Difference in Percentages = -2.6, 95% CI 2-sided [-8.5 to 3.4] — Differences in percentages of participants between groups and their 95% CIs were calculated based on MH proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)
Statistical Analysis 2: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.39, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

4. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 20 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 314 | 315
percentage of participants | 87.6 | 87.3
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; Difference in Percentages = 0.4, 95% CI 2-sided [-4.8 to 5.6] — The differences in percentages of participants between treatment groups and their 95% CIs were calculated based on the MH proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)
Statistical Analysis 2: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.87, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

5. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 20 Copies/mL at Week 96 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 314 | 315
percentage of participants | 83.4 | 84.8
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; Difference in Percentages = -1.2, 95% CI 2-sided [-6.9 to 4.6] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.69, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

6. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 20 Copies/mL at Week 144 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 144 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 144
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 314 | 315
percentage of participants | 78.0 | 82.2
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; Difference in Percentages = -4.2, 95% CI 2-sided [-10.5 to 2.1] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.19, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

7. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 295 | 302
log10 copies/mL | -3.11 (0.641) | -3.07 (0.738)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.48, ANOVA; p-value was adjusted by baseline HIV-1 RNA stratum and region stratum; Difference in LSM = -0.03, 95% CI 2-sided [-0.12 to 0.06] — Difference in least-squares mean (LSM), and its 95% confidence interval (CI) were adjusted by baseline HIV-1 RNA stratum and region stratum

8. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 279 | 288
log10 copies/mL | -3.09 (0.643) | -3.10 (0.705)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.99, ANOVA; Difference in LSM = 0.00, 95% CI 2-sided [-0.09 to 0.09] — Difference in LSM, and its 95% CI were adjusted by baseline HIV-1 RNA stratum and region stratum

9. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA at Week 144
Time Frame: Baseline, Week 144
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 260 | 269
log10 copies/mL | -3.11 (0.639) | -3.10 (0.681)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.88, ANOVA; Difference in LSM = 0.01, 95% CI 2-sided [-0.08 to 0.10] — Difference in LSM, and its 95% CI were adjusted by baseline HIV-1 RNA stratum and region stratum

10. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 294 | 300
cells/µL | 235 (185.8) | 228 (188.7)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.69, ANOVA; P-value was adjusted by the baseline HIV-1 RNA and region stratum; Difference in LSM = 6, 95% CI 2-sided [-24 to 36] — Difference in LSM, and its 95% CI were adjusted by the baseline HIV-1 RNA and region stratum

11. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 276 | 286
cells/µL | 287 (206.9) | 288 (246.8)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.94, ANOVA; P-value was adjusted by the baseline HIV-1 RNA and region stratum; Difference in LSM = -1, 95% CI 2-sided [-39 to 36] — Difference in LSM, and its 95% CI were adjusted by the baseline HIV-1 RNA and region stratum

12. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 144
Time Frame: Baseline, Week 144
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 255 | 260
cells/µL | 299 (224.9) | 317 (219.5)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.30, ANOVA; p-value was adjusted by baseline HIV-1 RNA stratum and region stratum; Difference in LSM = -20, 95% CI 2-sided [-59 to 18] — Difference in LSM, and its 95% CI were adjusted by baseline HIV-1 RNA stratum and region stratum

13. Secondary Outcome: Percentage Change From Baseline in Hip BMD at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 278 | 281
percentage change | -0.802 (2.3280) | -1.148 (2.5126)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.092, ANOVA; Difference in LSM = 0.346, 95% CI 2-sided [-0.057 to 0.748]

14. Secondary Outcome: Percentage Change From Baseline in Hip BMD at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 250 | 257
percentage change | -1.128 (2.7702) | -1.262 (2.8524)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.59, ANOVA; Difference in LSM = 0.135, 95% CI 2-sided [-0.356 to 0.625]

15. Secondary Outcome: Percentage Change From Baseline in Hip BMD at Week 144
Time Frame: Baseline, Week 144
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 236 | 240
percentage change | -1.020 (3.7638) | -1.291 (3.1140)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.39, ANOVA; Difference in LSM = 0.271, 95% CI 2-sided [-0.351 to 0.893]

16. Secondary Outcome: Percentage Change From Baseline in Spine BMD at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 284 | 285
percentage change | -0.772 (3.2228) | -0.552 (3.0956)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.41, ANOVA; Difference in LSM = -0.221, 95% CI 2-sided [-0.741 to 0.300]

17. Secondary Outcome: Percentage Change From Baseline in Spine BMD at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 256 | 258
percentage change | -0.705 (3.8721) | -0.219 (3.5159)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.14, ANOVA; Difference in LSM = -0.485, 95% CI 2-sided [-1.126 to 0.155]

18. Secondary Outcome: Percentage Change From Baseline in Spine BMD at Week 144
Time Frame: Baseline, Week 144
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 243 | 244
percentage change | -0.371 (4.4369) | 0.035 (3.5182)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.26, ANOVA; Difference in LSM = -0.406, 95% CI 2-sided [-1.119 to 0.307]

19. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 48 Open-Label as Defined by Missing = Excluded Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL was analyzed using Missing = Excluded for imputing missing HIV-1 RNA values using the All B/F/TAF Analysis Set. All missing data was excluded in the computation of the percentages (ie, missing data points were excluded from both the numerator and denominator in the computation). The denominator for percentages at a visit was the number of participants in the all B/F/TAF analysis set with non-missing HIV-1 RNA value at that visit.
Time Frame: Baseline, open-label Week 48
Population: Participants in All B/F/TAF Analysis Set (who were randomized into the randomized phase of the study and received at least 1 dose of the B/F/TAF in the randomized phase or at least 1 dose of the B/F/TAF in the open label extension phase) with available data were analyzed. For the B/F/TAF group, Week 48 open-label time point refers to Week 192; for Missing = Excluded analysis, it included the available participants at that time point from the Randomized Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All B/F/TAF: Blinded Phase: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) tablets fixed-dose combination (FDC) + abacavir (ABC)/dolutegravir (DTG)/lamivudine (3TC) (ABC/DTG/3TC) placebo orally once daily for at least 144 weeks, without regard to food.
  Open-Label Extension Phase: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive open-label (OL) B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
- ABC/DTG/3TC to B/F/TAF: Open Label Extension Phase: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive open-label (OL) B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
Arm/Group | All B/F/TAF | ABC/DTG/3TC to B/F/TAF
Number analyzed (Participants) | 237 | 212
percentage of participants | 99.2 [97.0 to 99.9] | 100 [98.3 to 100.0]

20. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 48 Open-Label as Defined by Missing = Failure Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL was analyzed using Missing = Failure for imputing missing HIV-1 RNA values using the All B/F/TAF Analysis Set. All missing data was treated as HIV-1 RNA ≥ 50 copies/mL. The denominator for percentages was the number of participants in all B/F/TAF analysis set.
Time Frame: Baseline, open-label Week 48
Population: Participants in the All B/F/TAF Analysis Set were analyzed. For the B/F/TAF group, Week 48 open-label time point refers to Week 192; for Missing = Failure analysis, it included all participants from the Randomized Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All B/F/TAF | ABC/DTG/3TC to B/F/TAF
Number analyzed (Participants) | 314 | 254
percentage of participants | 74.8 [69.7 to 79.5] | 83.5 [78.3 to 87.8]

21. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 96 Open-Label as Defined by Missing = Excluded Algorithm
Description: as for outcome 19
Time Frame: Baseline, open-label Week 96
Population: Participants in the All B/F/TAF Analysis Set with available data were analyzed. For the B/F/TAF group, Week 96 open-label time point refers to Week 240; for Missing = Excluded analysis, it included the available participants at that time point from the Randomized Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All B/F/TAF | ABC/DTG/3TC to B/F/TAF
Number analyzed (Participants) | 213 | 218
percentage of participants | 97.7 [94.6 to 99.2] | 99.5 [97.5 to 100.0]

22. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 96 Open-Label as Defined by Missing = Failure Algorithm
Description: as for outcome 20
Time Frame: Baseline, open-label Week 96
Population: Participants in the All B/F/TAF Analysis Set were analyzed. For the B/F/TAF group, Week 96 open-label time point refers to Week 240; for Missing = Failure analysis, it included all participants from the Randomized Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All B/F/TAF | ABC/DTG/3TC to B/F/TAF
Number analyzed (Participants) | 314 | 254
percentage of participants | 66.2 [60.7 to 71.5] | 85.4 [80.5 to 89.5]

23. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48 Open-Label
Time Frame: Baseline, open-label Week 48
Population: Participants in the All B/F/TAF Analysis Set with available data were analyzed. For the B/F/TAF group, Week 48 open-label time point refers to Week 192; for Change from Baseline in CD4 Cell Count analysis, it included the available participants at that time point from the Randomized Phase.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | All B/F/TAF | ABC/DTG/3TC to B/F/TAF
Number analyzed (Participants) | 234 | 212
cells/µL | 330 (242.8) | -4 (202.0)

24. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96 Open-Label
Time Frame: Baseline, open-label Week 96
Population: Participants in the All B/F/TAF Analysis Set with available data were analyzed. For the B/F/TAF group, Week 96 open-label time point refers to Week 240; for Change from Baseline in CD4 Cell Count analysis, it included the available participants at that time point from the Randomized Phase.
Measure: Mean (Standard Deviation); unit: cell/µL
Arm/Group | All B/F/TAF | ABC/DTG/3TC to B/F/TAF
Number analyzed (Participants) | 205 | 204
cell/µL | 339 (237.8) | -15 (188.1)

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose date (maximum: 279 weeks) plus 30 days All-Cause Mortality: Randomization date through last visit/follow up date (maximum duration: 282.4 weeks)
Description: Adverse Events: Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
  All-Cause Mortality: All Randomized Analysis Set included all participants randomized into the study.
Groups:
- B/F/TAF: B/F/TAF (50/200/25 mg) FDC tablet + ABC/DTG/3TC placebo orally once daily for at least 144 weeks, without regard to food.
- ABC/DTG/3TC: ABC/DTG/3TC (600/50/300 mg) FDC tablet + B/F/TAF placebo orally once daily for at least 144 weeks, without regard to food.
- B/F/TAF to B/F/TAF: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
Arm/Group | B/F/TAF | ABC/DTG/3TC | B/F/TAF to B/F/TAF | ABC/DTG/3TC to B/F/TAF
All-Cause Mortality (participants affected / at risk) | 2/316 | 1/315 | 2/252 | 2/254
Serious Adverse Events (participants affected / at risk) | 44/314 | 54/315 | 19/252 | 19/254
Other Adverse Events (participants affected / at risk) | 262/314 | 276/315 | 152/252 | 153/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=314) | ABC/DTG/3TC (N=315) | B/F/TAF to B/F/TAF (N=252) | ABC/DTG/3TC to B/F/TAF (N=254)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Middle ear adhesions (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Blindness transient (Eye disorders) | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Steatorrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 2 | 2 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 2 | 2 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 3 | 2 | 0 | 0
Appendicitis perforated (Infections and infestations) | 2 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 2
Complicated appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 2 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Fungaemia (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Gonococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Gonorrhoea (Infections and infestations) | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Injection site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 0 | 0
Neurosyphilis (Infections and infestations) | 1 | 2 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 | 0 | 0
Psychiatric evaluation (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Borderline personality disorder (Psychiatric disorders) | 1 | 1 | 0 | 0
Delirium tremens (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination, tactile (Psychiatric disorders) | 0 | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 3 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 3 | 1 | 1
Suicide attempt (Psychiatric disorders) | 2 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Endometrial thickening (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Penile necrosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alcohol use (Social circumstances) | 0 | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=314) | ABC/DTG/3TC (N=315) | B/F/TAF to B/F/TAF (N=252) | ABC/DTG/3TC to B/F/TAF (N=254)
Abdominal pain (Gastrointestinal disorders) | 18 | 23 | 5 | 6
Constipation (Gastrointestinal disorders) | 15 | 17 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 54 | 57 | 6 | 13
Nausea (Gastrointestinal disorders) | 40 | 77 | 8 | 7
Vomiting (Gastrointestinal disorders) | 18 | 24 | 3 | 7
Fatigue (General disorders) | 35 | 41 | 7 | 11
Pyrexia (General disorders) | 15 | 19 | 8 | 8
Seasonal allergy (Immune system disorders) | 7 | 16 | 3 | 5
Anal chlamydia infection (Infections and infestations) | 16 | 29 | 6 | 11
Bronchitis (Infections and infestations) | 20 | 30 | 3 | 2
Chlamydial infection (Infections and infestations) | 23 | 13 | 8 | 8
Covid-19 (Infections and infestations) | 0 | 0 | 20 | 23
Gastroenteritis (Infections and infestations) | 17 | 21 | 6 | 8
Gonorrhoea (Infections and infestations) | 22 | 21 | 5 | 5
Influenza (Infections and infestations) | 22 | 16 | 4 | 9
Nasopharyngitis (Infections and infestations) | 41 | 52 | 18 | 14
Pharyngitis (Infections and infestations) | 17 | 23 | 6 | 5
Proctitis gonococcal (Infections and infestations) | 17 | 21 | 9 | 13
Sinusitis (Infections and infestations) | 15 | 23 | 3 | 4
Syphilis (Infections and infestations) | 43 | 51 | 22 | 22
Upper respiratory tract infection (Infections and infestations) | 46 | 61 | 16 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 41 | 13 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 43 | 15 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 13 | 9 | 12
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 19 | 6 | 3
Dizziness (Nervous system disorders) | 10 | 19 | 2 | 2
Headache (Nervous system disorders) | 44 | 56 | 8 | 9
Anxiety (Psychiatric disorders) | 31 | 21 | 11 | 12
Depression (Psychiatric disorders) | 19 | 27 | 4 | 12
Insomnia (Psychiatric disorders) | 27 | 35 | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 22 | 13 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 35 | 13 | 6
Rash (Skin and subcutaneous tissue disorders) | 30 | 32 | 10 | 6
Hypertension (Vascular disorders) | 24 | 16 | 8 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (7):
  • Study Protocol: Original (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT02607930/Prot_004.pdf
  • Study Protocol: Amendment 1 (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT02607930/Prot_005.pdf
  • Study Protocol: Amendment 2 (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT02607930/Prot_006.pdf
  • Study Protocol: Amendment 3 (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT02607930/Prot_008.pdf
  • Statistical Analysis Plan: Original (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT02607930/SAP_007.pdf
  • Statistical Analysis Plan: Amendment 1 (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT02607930/SAP_009.pdf
  • Statistical Analysis Plan: Final Analysis (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT02607930/SAP_010.pdf